CLINICAL TRIAL: NCT04734821
Title: Prospective Study on the Contribution of Fluorescence in the Guidance of Lymphadenectomy and in Peroperative Evaluation of Pre-anastomotic Tissue Perfusion in Laparoscopic Esogastric Oncologic Resections
Brief Title: Fluorescence Image Guided Foregut Surgery
Acronym: FOREGUT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IHU Strasbourg (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 20-003
Record Dates: First submitted 2021-01-28; First posted 2021-02-02 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Esophageal Cancer; Gastric Cancer
Keywords: Esophageal cancer; Gastric cancer; Lymphadenectomy; Complications; Anastomosis
MeSH Terms: conditions — Esophageal Neoplasms; Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- NIR Fluorescence guided lymphadenectomy and anastomosis (Experimental)
  Interventions: Procedure: Near Infra-Red Fluorescence Guided Surgery

INTERVENTIONS:
Procedure: Near Infra-Red Fluorescence Guided Surgery — ICG injection around tumor each four direction by endoscopy followed by NIR fluorescence guidance laparoscopic or robotic esophagectomy or gastrectomy

SUMMARY:
A high number of resected lymph nodes is an independent prognostic factor for improved survival after esophagectomy or gastrectomy for cancer. The quality of the lymphadenectomy is operator-dependent, as is the evaluation of the vascularization of the digestive structures that are anastomosed to restore digestive continuity after esophago-gastric resection. The aim of the study is to evaluate the impact of Indocyanine Green (ICG) and near infra-red (NIR) fluorescence imaging guidance in terms of number of lymph nodes resected and quality of gastrointestinal tract anastomoses in esophagogastric cancer surgery.

DETAILED DESCRIPTION:
In cancer surgery, an oncological resection involves the resection of the primary lesion but also of the loco-regional lymph nodes.In the large retrospective study of the Global Group of esophageal cancer collaboration (WECC) involving 3,572 patients having had resection of the main tumor (60% adenocarcinomas, 40% squamous cell carcinomas), a high total number of resected lymph nodes has been shown to be an independent prognostic factor of improved survival after esophagectomy for esophageal or gastroesophageal junction cancer. The maximum survival at 5 years is modulated by the T classification: it is recommended to resect 10 lymph nodes for a "pT1" stage tumor (pathologic tumor stage 1), 20 for a "pT2" stage and at least 30 for a "pT3" / "T4" stage. This number is important in terms of staging, the decision of adjuvant treatments and prognostic. A recent European study showed that the average number of resected lymph nodes was 20. In addition, lymphatic drainage is variable according to the type and location of tumors, involving an adapted lymphadenectomy strategy to each situation.

Also in gastric cancer, a complete resection (R0) and adequate lymphadenectomy are predictive factors for healing and long-term survival. Lymphadenectomy is adapted to the type, stage and location of the primary lesion.

In the U.S., the National Cancer Network guidelines recommend a D2 lymphadenectomy or a minimum of 15 lymph nodes (Lymph Node, LN) recovered.However, most international guidelines consider the recovery of only 15 LNs is insufficient. A recent Korean study on more than 25,000 patients showed that the maximum survival advantage is observed by performing a lymphadenectomy with a minimum of 29 LNs recovered. The experience of Western surgeons is much less than that of surgeons in Asia, and it seems obvious that an intraoperative guidance method would be a major support for the decision making in real time and thus remove the current variability related to the level of experience of the surgeon.

In addition, oncology surgery includes in the vast majority of cases a resection of an segment of the digestive tract and requires the restoration of digestive continuity by simple anastomosis and/or by interposition of another intestinal segment.

This stage of the surgical procedure is critical, since any anastomotic leakage is burdened with a risk of complication sometimes lethal. The surgeon's experience, which allows him to evaluate visually the vascularization of the tissue to be anastomosed, is therefore fundamental to prevent the problems.

In esogastric surgery, anastomotic leaks are associated with increased postoperative morbidity, an extended stay in the Intensive Care Unit (ICU), a longer overall hospital stay,reduced quality of life and, in the context of cancer, shortened cancer-specific survival.

Several studies have identified risk factors for anastomotic leakage, such as chemoradiotherapy, surgical technique, smoking, diabetes, and the location of the anastomosis. These factors may compromise the perfusion of the replacement conduit after esophagectomy and gastrectomy and increase the risk of anastomotic leakage. Objective assessment of tissue perfusion could be an excellent tool to identify ischemia of the conduits and thus reduce the incidence of anastomotic leaks. A perfusion compromise of the proximal portion of the gastric conduit, used for the recovery of the digestive continuity after esophagectomy, has been identified as one of the risk factors of digestive fistula.

It is therefore obvious that at the present time, for curative cancer resection or reconstruction after esogastric resection surgery, the outcome of the treatment depends mainly on the surgeon's experience and perception of the surgical field.

Today, the development of specific fluorescence imaging devices enables the surgeons to visualize tumors and vascular and lymphatic structures. This technology is expected to increase the reproducibility of esogastric surgery and its results.

The proposed study is based on the hypothesis that Fluorescence Image Guided Surgery (FIGS) would improve the quality and reproducibility of esophageal and stomach oncology surgery (lymphadenectomy and complete resection), as well as to decrease the risk of anastomotic complications after resective surgery of the esophagus or part or all of the stomach (study of the vascularization).

ELIGIBILITY:
Inclusion Criteria:

* Man or woman over 18 years old.
* Patient with resectable primitive esophageal or gastric cancer confirmed by biopsy without distant metastases
* Patient with no contraindications to anaesthesia and performance of esophageal and/or gastric surgery
* Patient able to receive and understand information related to the study and give written informed consent.
* Patient affiliated to the French social security system.

Exclusion Criteria:

* Patient undergoing emergency surgery (hemorrhage, occlusion or perforation).
* Presence of distant metastasis
* Patient at risk of allergy to indocyanine green or to other fluorescent compounds
* Pregnant or lactating patient.
* Patient in exclusion period (determined by a previous or a current study).
* Patient under the protection of justice.
* Patient under guardianship or trusteeship.
* Patient deprived of liberty

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the usefulness of ICG fluorescence to guide lymphadenectomy in oncological esogastric resections | During the surgical procedure
  Additional detection (YES-NO) of lymph nodes after activation of the NIR fluorescence guidance system during lymphadenectomy.

SECONDARY OUTCOMES:
Evaluation of the impact of fluorescence guidance on the number of resected lymph nodes in oncological esogastric resections | 7 days after operation when pathologic result was reported
  Number of lymph nodes, counted in anatomopathological analysis, obtained after fluorescence-guided lymphadenectomy in the esogastric oncology resections compared to historical data
Evaluation of the impact of fluorescence guidance in intraoperative evaluation of pre-anastomotic tissue perfusion | 30 days after operation
  Anastomotic fistula rate after fluorescence control of pre-anastomotic vascularisation in oncological esogastric resections compared to historical data

CONTACTS AND LOCATIONS:
Overall Officials: Silvana PERRETTA, MD, PhD, Principal Investigator — Service de Chirurgie Digestive et Endocrinienne, NHC, Strasbourg
Locations (1):
- Service de Chirurgie Digestive et Endocrinienne, NHC, Strasbourg, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rosenthal EL, Warram JM, Bland KI, Zinn KR. The status of contemporary image-guided modalities in oncologic surgery. Ann Surg. 2015 Jan;261(1):46-55. doi: 10.1097/SLA.0000000000000622. PMID 25599326
- [Background] van der Werf LR, Dikken JL, van Berge Henegouwen MI, Lemmens VEPP, Nieuwenhuijzen GAP, Wijnhoven BPL; Dutch Upper GI Cancer Audit group. A Population-based Study on Lymph Node Retrieval in Patients with Esophageal Cancer: Results from the Dutch Upper Gastrointestinal Cancer Audit. Ann Surg Oncol. 2018 May;25(5):1211-1220. doi: 10.1245/s10434-018-6396-7. Epub 2018 Mar 9. PMID 29524046
- [Background] Tachimori Y. Pattern of lymph node metastases of squamous cell esophageal cancer based on the anatomical lymphatic drainage system: efficacy of lymph node dissection according to tumor location. J Thorac Dis. 2017 Jul;9(Suppl 8):S724-S730. doi: 10.21037/jtd.2017.06.19. PMID 28815068
- [Background] Nafteux P, Depypere L, Van Veer H, Coosemans W, Lerut T. Principles of esophageal cancer surgery, including surgical approaches and optimal node dissection (2- vs. 3-field). Ann Cardiothorac Surg. 2017 Mar;6(2):152-158. doi: 10.21037/acs.2017.03.04. PMID 28447004
- [Background] Songun I, Putter H, Kranenbarg EM, Sasako M, van de Velde CJ. Surgical treatment of gastric cancer: 15-year follow-up results of the randomised nationwide Dutch D1D2 trial. Lancet Oncol. 2010 May;11(5):439-49. doi: 10.1016/S1470-2045(10)70070-X. Epub 2010 Apr 19. PMID 20409751
- [Background] Woo Y, Goldner B, Ituarte P, Lee B, Melstrom L, Son T, Noh SH, Fong Y, Hyung WJ. Lymphadenectomy with Optimum of 29 Lymph Nodes Retrieved Associated with Improved Survival in Advanced Gastric Cancer: A 25,000-Patient International Database Study. J Am Coll Surg. 2017 Apr;224(4):546-555. doi: 10.1016/j.jamcollsurg.2016.12.015. Epub 2016 Dec 23. PMID 28017807
- [Background] Vahrmeijer AL, Hutteman M, van der Vorst JR, van de Velde CJ, Frangioni JV. Image-guided cancer surgery using near-infrared fluorescence. Nat Rev Clin Oncol. 2013 Sep;10(9):507-18. doi: 10.1038/nrclinonc.2013.123. Epub 2013 Jul 23. PMID 23881033
- [Background] Herrera-Almario G, Patane M, Sarkaria I, Strong VE. Initial report of near-infrared fluorescence imaging as an intraoperative adjunct for lymph node harvesting during robot-assisted laparoscopic gastrectomy. J Surg Oncol. 2016 Jun;113(7):768-70. doi: 10.1002/jso.24226. Epub 2016 Mar 29. PMID 27021142
- [Background] Kwon IG, Son T, Kim HI, Hyung WJ. Fluorescent Lymphography-Guided Lymphadenectomy During Robotic Radical Gastrectomy for Gastric Cancer. JAMA Surg. 2019 Feb 1;154(2):150-158. doi: 10.1001/jamasurg.2018.4267. PMID 30427990
- [Background] Kim TH, Kong SH, Park JH, Son YG, Huh YJ, Suh YS, Lee HJ, Yang HK. Assessment of the Completeness of Lymph Node Dissection Using Near-infrared Imaging with Indocyanine Green in Laparoscopic Gastrectomy for Gastric Cancer. J Gastric Cancer. 2018 Jun;18(2):161-171. doi: 10.5230/jgc.2018.18.e19. Epub 2018 Jun 28. PMID 29984066
- [Background] Turner SR, Molena DR. The Role of Intraoperative Fluorescence Imaging During Esophagectomy. Thorac Surg Clin. 2018 Nov;28(4):567-571. doi: 10.1016/j.thorsurg.2018.07.009. PMID 30268302
- [Background] Hachey KJ, Gilmore DM, Armstrong KW, Harris SE, Hornick JL, Colson YL, Wee JO. Safety and feasibility of near-infrared image-guided lymphatic mapping of regional lymph nodes in esophageal cancer. J Thorac Cardiovasc Surg. 2016 Aug;152(2):546-54. doi: 10.1016/j.jtcvs.2016.04.025. Epub 2016 Apr 11. PMID 27179838
- [Background] Park SY, Suh JW, Kim DJ, Park JC, Kim EH, Lee CY, Lee JG, Paik HC, Chung KY. Near-Infrared Lymphatic Mapping of the Recurrent Laryngeal Nerve Nodes in T1 Esophageal Cancer. Ann Thorac Surg. 2018 Jun;105(6):1613-1620. doi: 10.1016/j.athoracsur.2018.01.083. Epub 2018 Mar 5. PMID 29518388
- [Background] Kaburagi T, Takeuchi H, Oyama T, Nakamura R, Takahashi T, Wada N, Saikawa Y, Kamiya S, Tanaka M, Wada T, Kitagawa Y. Intraoperative fluorescence lymphography using indocyanine green in a patient with chylothorax after esophagectomy: report of a case. Surg Today. 2013 Feb;43(2):206-10. doi: 10.1007/s00595-012-0391-6. Epub 2012 Oct 30. PMID 23108512
- [Background] Kim M, Son SY, Cui LH, Shin HJ, Hur H, Han SU. Real-time Vessel Navigation Using Indocyanine Green Fluorescence during Robotic or Laparoscopic Gastrectomy for Gastric Cancer. J Gastric Cancer. 2017 Jun;17(2):145-153. doi: 10.5230/jgc.2017.17.e17. Epub 2017 Jun 9. PMID 28680719
- [Background] Zehetner J, DeMeester SR, Alicuben ET, Oh DS, Lipham JC, Hagen JA, DeMeester TR. Intraoperative Assessment of Perfusion of the Gastric Graft and Correlation With Anastomotic Leaks After Esophagectomy. Ann Surg. 2015 Jul;262(1):74-8. doi: 10.1097/SLA.0000000000000811. PMID 25029436
- [Background] Campbell C, Reames MK, Robinson M, Symanowski J, Salo JC. Conduit Vascular Evaluation is Associated with Reduction in Anastomotic Leak After Esophagectomy. J Gastrointest Surg. 2015 May;19(5):806-12. doi: 10.1007/s11605-015-2794-3. Epub 2015 Mar 20. PMID 25791907
- [Background] Agzarian J, Visscher SL, Knight AW, Allen MS, Cassivi SD, Nichols FC 3rd, Shen KR, Wigle D, Blackmon SH. The cost burden of clinically significant esophageal anastomotic leaks-a steep price to pay. J Thorac Cardiovasc Surg. 2019 May;157(5):2086-2092. doi: 10.1016/j.jtcvs.2018.10.137. Epub 2018 Nov 15. PMID 30558876
- [Background] Carrott PW, Markar SR, Kuppusamy MK, Traverso LW, Low DE. Accordion severity grading system: assessment of relationship between costs, length of hospital stay, and survival in patients with complications after esophagectomy for cancer. J Am Coll Surg. 2012 Sep;215(3):331-6. doi: 10.1016/j.jamcollsurg.2012.04.030. Epub 2012 Jun 8. PMID 22683069
- [Background] Wang S, Xu L, Wang Q, Li J, Bai B, Li Z, Wu X, Yu P, Li X, Yin J. Postoperative complications and prognosis after radical gastrectomy for gastric cancer: a systematic review and meta-analysis of observational studies. World J Surg Oncol. 2019 Mar 18;17(1):52. doi: 10.1186/s12957-019-1593-9. PMID 30885211
- [Background] Carus T, Dammer R. Laparoscop fluorescence angiography with indocyanine green to control the perfusion of gastrointestinal anastomoses intraoperatively. Surg Technol Int. 2012 Dec;22:27-32. PMID 23315721